CLINICAL TRIAL: NCT05160220
Title: Double-blind Placebo-controlled Naturalistic Study of Microdosing With Psilocybin: Effects on Brain Activity, Behavior, Cognition, Creativity, and Mental Health
Brief Title: Naturalistic Study of Microdosing With Psilocybin
Acronym: NATMICRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Council of Scientific and Technical Research, Argentina (Other Government)
Responsible Party: Principal Investigator, Enzo Tagliazucchi, Principal Investigator, National Council of Scientific and Technical Research, Argentina
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 001
Record Dates: First submitted 2021-05-05; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Cognitive Change; Creativity; Mood Change; Sleep
Keywords: psilocybin; psychedelics; nootropics; microdosing; EEG; cognition; creativity; behavior; sleep
MeSH Terms: conditions — Behavior | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psilocybe cubensis (Active Comparator): 0.5 g dried and powdered P. cubensis in gel capsules, dosing on two separate days, separated by one week from the placebo, randomized order.
  Interventions: Drug: Psilocybin
- Inactive placebo (Placebo Comparator): Same weight of inactive placebo in gel capsules, dosing on two separate days, separated by one week from the placebo, randomized order.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Psilocybin — 0.5 g dried Psilocybe cubensis mushroom material, 0.8 mg psilocybin.
  Arms: Psilocybe cubensis
Drug: Placebo — 0.5 g dried edible non-psychoactive mushroom material.
  Arms: Inactive placebo

SUMMARY:
This study seeks to understand the neural, cognitive and behavioral effects of low doses of psilocybin administered in the form of dried mushroom material (0.5 g of Psilocybe cubensis) consumed in natural settings following a placebo-controlled double-blind experimental design.

DETAILED DESCRIPTION:
Sub-threshold doses of serotonergic psychedelics are frequently consumed as cognitive enhancers, and due to their purported positive effects on mood, energy and creativity ("microdosing").

The acute and short-term effects of psilocybin (the psychoactive compound of Psilocybe cubensis mushrooms) on several variables will be investigated, comprising spontaneous and evoked electrophysiological brain activity, perception and cognitive function (cognitive flexibility, attention, inhibitory control, conscious access, visual perception), creativity (problem solving, divergent and convergent thinking), behavior (actigraphy and sleep patterns, natural language production) and several domains related to well-being and mental health of the participants.

This study is simultaneously naturalistic (i.e. recruited subjects are intrinsically motivated to microdose, as they have decided to embark in a microdosing protocol) and controlled by expectations, following a double-blind placebo-controlled design. Participants will microdose according to the following schedule:

Two sessions (0.5 g dried Psilocybin mushrooms vs. dried edible mushroom material without psychoactive effects as a placebo condition) will be conducted. A third party will be in charge of generating their active dose and placebo capsules, and they will also implement a blinding procedure.

Each session will span one week of measurements. Subjects will be given a smartwatch to monitor activity and sleeping patterns at the beginning of the week. At days 3 and 5, subjects will take capsules with active mushroom material or placebo, and then several variables will be recorded. Experiments will be conducted in a setting that is natural and comfortable for the participants, e.g. their homes.

The main outcome measures consist of resting state activity recorded with EEG, evoked response potentials and performance during cognitive tasks, behavioral variables obtained with actigraphy and automated sleep scoring, natural language analysis, and several measurs self-reported via standarized questionnaires.

After completion, this study will provide direct evidence concerning the efficacy of microdosing for cognitive enhancement under natural conditions, i.e. those most frequently used by individuals who microdose, as well as provide information concerning the potential underlying neurobiological mechanisms.

ELIGIBILITY:
Inclusion Criteria:

1. Men and woman with more than 21 years.
2. Participans are planning to microdose using their own dried mushroom material and adhere to the experimental protocol.
3. No active psychiatric conditions requiring treatment with psychotropic medications.
4. Able to provide informed consent.

Excusion Criteria:

1. Use of psychotropic medication during the study, including stimulants such as caffeine.
2. Prior adverse reactions to psychedelics according to the Challenging Experiences Questionnaire administered during initial screening.
3. Pregnant women or women during lactation
4. History of high or low blood pressure or other cardiovascular risks.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Resting state oscillations measured with EEG | 1 week
  Our goal is to study changes in spectral content before and during the acute effects with the purpose of comparing changes with those observed under higher doses of psilocybin.
Attention | 1 week
  Measured performance in the attentional blink paradigm
Inhibitory control | 1 week
  Measured using the go/no go experimental paradigm
Conscious access | 1 week
  Measured using the backward masking paradigm
Visual perception | 1 week
  Measured using the binocular rivalry paradigm
Physical activity | 1 week
  Measured using wrist actigraphy using a smartwach
Divergent thinking | 1 week
  Measured using the Alternative Uses Task (AUT)
Attention | 1 week
  Measured using the hiearchical mismatch negativity paradigm combined with EEG
Cognitive flexibility | 1 week
  Measured using the stroop task
Convergent thinking | 1 week
  Measured using the Remote Associations Task (RAT)
Convergent thinking | 1 week
  Measured using the Wallach-Kogan test (WK)

SECONDARY OUTCOMES:
Effect positive/negative affect and well-being | 1 week
  Measured using the Positive and Negative Affect Schedule (PANAS)
Effects on anxiety | 1 week
  Measured using State Trait Anxiety Inventory (STAI)
Effects on personality | 1 week
  Measured using the Big Five inventory (BFI)
Concentration of psilocybin in the dried material | 1 week
  To be measured using high performance liquid chromatography

CONTACTS AND LOCATIONS:
Overall Officials: Enzo Tagliazucchi, PhD, Principal Investigator — National Council of Scientific and Technical Research, Argentina
Locations (1):
- Instituto de Fisica de Buenos Aires (IFIBA), Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
All raw data will be made available online through a data sharing webside (e.g. Zenodo) upon publication of the pre-pring containing the results of our study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication, indefinite.
Access Criteria: Public
URL: https://zenodo.org/